CLINICAL TRIAL: NCT06068036
Title: Telehealth Intervention Involving the HEARTS Technical Package and the Use of an Activity Monitor to Increase Physical Activity Level Post-stroke: a Feasibility Randomized Controlled Trial
Brief Title: Telehealth Intervention Involving HEARTS Technical Package and Activity Monitor to Promote Physical Activity Post-stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Minas Gerais (Other)
Collaborators: Fundação de Amparo à Pesquisa do estado de Minas Gerais (Other); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government); Coordenaçao de Aperfeiçoamento de Pessoal de Nível Superior (Unknown); Worldwide Universities Network (Unknown)
Responsible Party: Principal Investigator, Christina Danielli Coelho de Morais Faria, Doctor, Federal University of Minas Gerais
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CAAE: 66980723.2.0000.5149
Record Dates: First submitted 2023-09-27; First posted 2023-10-05 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Stroke
Keywords: Stroke; Physical activity; Telehealth; Feasibility Study; Randomized controlled trial
MeSH Terms: conditions — Stroke; Motor Activity | interventions — Fitness Trackers

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The collection will be performed by a previously trained examiner, blinded to the allocation of groups. All participants will be instructed not to comment on information about the training received. All statistical analyzes will be performed by an independent examiner, blinded to all procedures performed in the study, including with regard to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental): Telehealth intervention involving the HEARTS technical package and the use of Smartwatch Mi Band 7® activity monitor. The HEARTS technical package presents the 5As brief intervention (Ask, Advise, Assess, Assist, Arrange) to promote physical activity participation. Participants will receive a physical activity monitor (as instructed in the HEARTS technical package) and will be monitored by telephone call, once a week, in order to reinforce successes and identify solutions to difficulties (as instructed in the HEARTS technical package) to practice physical activity. These individuals will undertake a 12-week intervention program. In the first week, individuals will perform the first four steps of the 5As brief intervention in person, where they will be instructed on how to use the physical activity monitor, they will receive a diary of regular physical activity practice, will be guided on how to fill it out, and will schedule the best times to receive the weekly telephone call.
  Interventions: Behavioral: Telehealth intervention: HEARTS technical package + activity monitor (Smartwatch Mi Band 7®)
- Control group (Active Comparator): Participants will undergo the same intervention as the experimental group, but will not receive the physical activity monitor (Smartwatch Mi Band 7®).
  Interventions: Behavioral: Telehealth intervention: HEARTS technical package

INTERVENTIONS:
Behavioral: Telehealth intervention: HEARTS technical package + activity monitor (Smartwatch Mi Band 7®) — Telehealth intervention involving the HEARTS technical package and the use of Smartwatch Mi Band 7® activity monitor. The HEARTS technical package presents the 5As brief intervention (Ask, Advise, Assess, Assist, Arrange) to promote physical activity participation. Participants will receive a physical activity monitor (as instructed in the HEARTS technical package) and will be monitored by telephone call, once a week, in order to reinforce successes and identify solutions to difficulties (as instructed in the HEARTS technical package) to practice physical activity. These individuals will undertake a 12-week intervention program. In the first week, individuals will perform the first four steps of the 5As brief intervention in person, where they will be instructed on how to use the physical activity monitor, they will receive a diary of regular physical activity practice, will be guided on how to fill it out, and will schedule the best times to receive the weekly telephone call.
  Arms: Experimental group
Behavioral: Telehealth intervention: HEARTS technical package — The same intervention as the experimental group, but without the additional use of the physical activity monitor (Smartwatch Mi Band 7®).
  Arms: Control group

SUMMARY:
Objectives: The aim of this feasibility randomized controlled trial (RCT) study is to investigate whether the theoretically informed telehealth intervention involving the HEARTS Technical Package and the use of an activity monitor to increase physical activity level post-stroke is feasible and to estimate the parameters for conducting a fully powered RCT.

Design: A Phase 1 feasibility RCT study with blinded assessment will assign eligible participants to experimental or control group. Participants in both groups will undergo a theoretically informed telehealth intervention based on the HEARTS technical package (a face-to-face session and telephone call follow-up). The experimental group will have additional use of the Mi Band 7® Smartwatch activity monitor. For both groups, the intervention will last for 12 weeks. The feasibility outcomes will be identified considering the different phases of conducting the study. A trained researcher, blinded to the group allocation, will collect the sociodemographic, anthropometric, and clinical outcomes, in a university laboratory setting.

Study Outcomes: Feasibility of recruitment, intervention, and measurement, and clinical outcomes.

Conclusions: Results from this feasibility RCT study will inform on the design and sample required for a fully powered RCT with a similar aim.

DETAILED DESCRIPTION:
Standard Operating Procedures: A non-probabilistic sample will be recruited from the community. Recruitment strategies include: referrals (e.g, phone numbers obtained from other research projects and university extension programs) and advertisements (e.g. physical folders distributed in public places, and electronic pamphlets published on social media). All subjects will be informed about the study procedures and will provide written consent. The feasibility outcomes will be identified considering the different phases of conducting the study. A trained researcher, blinded to the group allocation, will collect the sociodemographic, anthropometric, and clinical outcomes, in a university laboratory setting. Two independent examiners, blinded to the group allocation, will enter the data into a statistical software package, verify any missing or apparently wrong values. Original paper forms will be kept in a secure place. Electronic files will be available only to the research team. Analysis will be carried-out by a researcher, blinded to the group allocation. All individuals will receive an identification code to ensure anonymity.

Statistical analyzes: All analyzes will be performed using SPSS (SPSS Inc., Chicago, IL, USA). Descriptive statistics will be calculated for all outcomes. The effect sizes will be calculated to determine the magnitude of within-groups and between-groups comparisons. The level of significance will be set at 5% and adjusted for multiple comparisons.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of stroke for more than six months;
* ≥18 years of age;
* Be rated as "Inactive" according to Human Activity Profile (HAP);
* Provide medical approval to practice physical activity.

Exclusion Criteria:

* Positive screening test for possible cognitive alterations;
* Pain or other adverse health condition that compromises the performance of the proposed intervention program, such as vestibular disorders, severe arthritis or any other diagnosis of disease of the nervous system.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-09-27 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Feasibility of recruitment | At enrolment and allocation.
  It will be determined by the ratio between the total number of eligible individuals (EI) and the total number of screened individuals (SI) (measure=EI/IS), and by the ratio between the total number of eligible individuals (EI) and the total number of recruited individuals (RI) (measure=EI/RI).
Feasibility of intervention (retention) | At allocation and post-intervention (week-12).
  It will be determined by the ratio between the total number of individuals who completed the proposed intervention program and the total number of individuals who started the proposed intervention program.
Feasibility of intervention (follow-up of individuals) | At allocation, post-intervention (week-12), and one month after the end of the intervention (week-16).
  It will be determined the ratio between the total number of individuals who remained in the same group to which they were initially allocated until follow-up and the total number of individuals who were allocated.
Feasibility of intervention (attendance) | At allocation and post-intervention (week-12).
  It will be determined by the ratio between the total number of sessions performed and the total number of sessions offered.
Feasibility of intervention (safety) | During the intervention (12 weeks) and follow-up (4 weeks).
  It will be determined by the number and reasons of adverse events (e.g. pain, falls, hospitalization, and death) identified during the period of intervention and follow-up of the individual.
Feasibility of intervention (perceived effectiveness) | At post-intervention (week-12).
  It will be determined by the following question: "Comparing how it was before you carried out the intervention and now, do you think that your ability to perform routine physical activity is: much worse, moderately worse, a little worse, the same, a little better, moderately better, or very better?".
Feasibility of measurement | At baseline, post-intervention (week-12), and one month after the end of the intervention (week-16).
  It will be determined by the percentage of clinical outcomes measured (ratio between the number of clinical outcomes measured and the number of clinical outcomes proposed to be measured), and the percentage of participants who filled-out the diary (ratio between the number of individuals who filled-out the diary and the number of individuals who started the proposed intervention program).

SECONDARY OUTCOMES:
Physical activity level | At baseline, post-intervention (week-12), and one month after the end of the intervention (week-16).
  Human Activity Profile (HAP). One of the outcomes provided by the instrument is the Maximum Activity Score (MAS). From the MAS, the Adjusted Activity Score (AAS) can be found by subtracting from the MAS the number of activities that the individual provided as the answer "I stopped doing". Higher scores indicate better outcome.
Number of post-stroke individuals who became physically active | At baseline, post-intervention (week-12), and one month after the end of the intervention (week-16).
  Human Activity Profile (HAP). One of the measures provided by the questionnaire is the "Activity Rating", which provides an overall rating of the respondent's activity level into "Inactive", "Moderately active" and "Active".
Systolic and diastolic blood pressure | At baseline, post-intervention (week-12), and one month after the end of the intervention (week-16).
  Tycos® aneroid sphygmomanometer (WelchAllyn Inc., NY, USA, Model DS44) and stethoscope (Litmann Classic II SE 3M®, USA).
Lifestyle-related energy consumption | At baseline, post-intervention (week-12), and one month after the end of the intervention (week-16).
  Human Activity Profile (HAP). One of the measures provided by the questionnaire is the "Lifestyle-related energy consumption", which provides a measure of actual oxygen consumption estimated from the "Activity Adjusted Score" (AAS). This measure is operationalized in ml.kg-1.min-1. Higher scores indicate better outcome.
Self-efficacy for physical activity | At baseline, post-intervention (week-12), and one month after the end of the intervention (week-16).
  Self-efficacy for Physical Activity Scale. The scale has 10 items and has two response options: "Yes" is computed as 1 and "No" is computed as 0. The total score is defined by the sum of the scores for each item. The minimum total score is 0 and the maximum total score is 10. The higher the total score, the higher the self-efficacy for physical activity.
Health-related quality of life | At baseline, post-intervention (week-12), and one month after the end of the intervention (week-16).
  Stroke Specific Quality of Life Scale (SS-QOL). The scale has 49 items across 12 domains (items are rated on a 5-point Likert scale) and has three different sets of responses (indicated on the scale). The total score is defined by the sum of the scores for each item. The minimum total score is 49 and the maximum total score is 245. The higher the total score, the better the health-related quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Christina Faria, PhD, Principal Investigator — Federal University of Minas Gerais
Locations (1):
- Universidade Federal de Minas Gerais, Belo Horizonte, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gladstone DJ, Lindsay MP, Douketis J, Smith EE, Dowlatshahi D, Wein T, Bourgoin A, Cox J, Falconer JB, Graham BR, Labrie M, McDonald L, Mandzia J, Ngui D, Pageau P, Rodgerson A, Semchuk W, Tebbutt T, Tuchak C, van Gaal S, Villaluna K, Foley N, Coutts S, Mountain A, Gubitz G, Udell JA, McGuff R, Heran MKS, Lavoie P, Poppe AY; Canadian Stroke Consortium. Canadian Stroke Best Practice Recommendations: Secondary Prevention of Stroke Update 2020. Can J Neurol Sci. 2022 May;49(3):315-337. doi: 10.1017/cjn.2021.127. Epub 2021 Jun 18. PMID 34140063
- [Background] Kleindorfer DO, Towfighi A, Chaturvedi S, Cockroft KM, Gutierrez J, Lombardi-Hill D, Kamel H, Kernan WN, Kittner SJ, Leira EC, Lennon O, Meschia JF, Nguyen TN, Pollak PM, Santangeli P, Sharrief AZ, Smith SC Jr, Turan TN, Williams LS. 2021 Guideline for the Prevention of Stroke in Patients With Stroke and Transient Ischemic Attack: A Guideline From the American Heart Association/American Stroke Association. Stroke. 2021 Jul;52(7):e364-e467. doi: 10.1161/STR.0000000000000375. Epub 2021 May 24. No abstract available. PMID 34024117
- [Background] Abe H, Orita M, Arichi S. Erythrocyte deformability in aging. Mech Ageing Dev. 1984 Oct 31;27(3):383-90. doi: 10.1016/0047-6374(84)90060-5. PMID 6513611
- [Background] Eldridge SM, Lancaster GA, Campbell MJ, Thabane L, Hopewell S, Coleman CL, Bond CM. Defining Feasibility and Pilot Studies in Preparation for Randomised Controlled Trials: Development of a Conceptual Framework. PLoS One. 2016 Mar 15;11(3):e0150205. doi: 10.1371/journal.pone.0150205. eCollection 2016. PMID 26978655
- [Derived] Peniche PDC, Lennon O, Magalhaes JP, Dos Santos JM, Polese JC, Faria CDCM. Telehealth intervention involving the HEARTS Technical Package and the additional use of an activity monitor to increase physical activity level post-stroke: Protocol for a feasibility randomized controlled trial. PLoS One. 2025 Apr 4;20(4):e0320026. doi: 10.1371/journal.pone.0320026. eCollection 2025. PMID 40184417